CLINICAL TRIAL: NCT07041437
Title: Efficacy and Safety Study of SHR-A2102-based Treatment in Advanced Breast Cancer
Brief Title: Study of SHR-A2102 Combined Other Antitumor Drugs in Advanced Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Hongxia Wang, Chief physician, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC-MUL-IIT-SHRA2102
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Advanced Breast Cancer

STUDY DESIGN:
Intervention Model Description: Two arms of SHR-A2102 based-treatment will be enrolled to evaluate efficacy and safety, but this is a nonrandomized design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-A2102 (Experimental): Single Agent
  Interventions: Drug: SHR-A2102
- SHR-A2102+adebrelimab (Experimental): SHR-A2102 combined with adebrelimab
  Interventions: Drug: SHR-A2102; Drug: Adebrelimab

INTERVENTIONS:
Drug: SHR-A2102 — ADC
Drug: Adebrelimab — PD-L1 inhibitor
  Arms: SHR-A2102+adebrelimab

SUMMARY:
Our study is aimed to evaluate the efficacy and safety of SHR-A2102 combined other antitumor treatments in advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 75 years old (including boundary values), patients with advanced or metastatic breast cancer;
* ECOG PS Score: 0~1;
* Based on RECIST v1.1, at least one measurable lesion;
* Patients must have a life expectancy ≥ 3 months;
* Adequate organ function and marrow function (no corrective treatment within 14 days before first dose);
* Women of childbearing potential (WOCBP) should agree to use an effective method of contraception and no lactation from the initiation of screening to 7 months after the last dose of study therapy; WOCBP should have a negative serum pregnancy result within 7 days before the first dose of study therapy; if unneutered male subjects (including using other sterilization except bilateral orchidectomy [e.g. vasectomy]) are willing to have sexual behaviour with WOCBP, one kind of contraception must be used to prevent the pregnancy of his partner from the date of enrolment to 7 months after the last dose of study therapy);
* Willing and able to provide written informed consent and comply with the requirements and restrictions in the protocol.

Exclusion Criteria:

* Active brain metastasis; Stable brain metastasis (at least 4 weeks after intracranial local treatment, subjects should meet one of the following requirements: a. no signs of disease progression confirmed by imaging; b. no clinical symptom, and not necessary to corticosteroid or anticonvulsant therapy; c. with clinical symptom, but not necessary to increase dose of corticosteroid or combine with dexamethasone to control clinical symptom compared with intracranial local treatment) is allowed to be enrolled;
* Existence of third space fluid (e.g. massive ascites, pleural effusion, pericardial effusion which needs drainage again to relieve symptoms within 4 weeks after the first drainage) which is not well controlled by effective methods, e.g. drainage;
* Other malignancy within prior 2 years with no necessary treatment (except hormone replacement treatment) for at least recent 2 years, except: curatively treated in situ cancer of the cervix, skin basal cell carcinoma, skin squamous cell carcinoma or papillary thyroid carcinoma;
* Has received antitumor surgery, radiotherapy, chemotherapy, targeted therapy or immunological therapy within 4 weeks before first dose of study therapy; has received antitumor endocrine therapy within one week before first dose of study therapy;
* Adverse events caused by prior antitumor therapy have not recovered to ≤grade 1 per NCI-CTCAE v5.0 (except alopecia and tolerable, chronic grade 2 toxicity determined by investigator);
* Use of other antitumor systemic treatment during the study;
* Has received CYP3A4, CYP2D6, P-gp or BCRP potent inhibitors or inducers <5-fold half-life of the drug before the first dose;
* Hypersensitivity to study therapy or any of its excipients;
* Has known clinically significant lung disease, including but not limited to: interstitial lung disease, pneumonitis, pulmonary fibrosis;
* Known history of immunodeficiency, including HIV-positive, other acquired or innate immunodeficient disease, or known history of organ transplantation, or known history of allogenic haemopoietic stem cell transplantation;
* Has active hepatitis B (HBsAg-positive and HBV DNA≥500 IU/mL), hepatitis C (positive for HCV antibody and HCV RNA above ULN) and hepatic cirrhosis;
* Has an active infection requiring antibiotics, antiviral or antifungal treatment, or pyrexia >38.5℃ of unknown origin during the screening period before first dose of study therapy (patients with pyrexia due to cancer could be enrolled determined by investigator);
* Known severe cardiac-cerebral vascular disease, including but not limited to: a) known severe cardiac rhythm or conduction disorder, such as ventricular arrhythmias necessary for clinical intervention, second or third degree atrioventricular block; b) under the resting state, QTcF>470ms for female or 450ms for male examined by 12-lead ECG; c) acute coronary syndrome, congestive heart failure (NYHA classification of heart failure ≥ Class II), myocardial infarction, aortic dissection, cerebral stroke, or other ≥grade 3 cardiac-cerebral vascular events; d) LVEF<50%; e) clinically uncontrolled hypertension;
* Existence of arterial/venous thrombotic event within 6 months before first dose, such as cerebrovascular accidents (including transient ischemic attack, cerebral haemorrhage and cerebral infarction), deep venous thrombosis and pulmonary embolism;
* (Arm 2 only) Has received or been receiving PD-1/PD-L1 inhibitor;
* (Arm 2 only) Has active autoimmune disease or a history of autoimmune disease (including but not limited to: autoimmune hepatitis, uveitis, inflammatory bowel disease, hypophysitis, vasculitis, nephritis, hyperthyroidism, uncontrolled hypothyroidism only treated with hormone replacement therapy); subject that has skin disease unnecessary for systemic treatment (such as vitiligo, psoriasis, alopecia), controlled type I diabetes treated with insulin, or complete remission of asthma in childhood and no need to any intervention in adulthood can be enrolled; subject that has asthma which needs medical intervention by bronchodilators can not be enrolled; subject that has been receiving chronic, systemic steroid therapy (daily dose >10mg prednisone or equivalent) or any other type of immunosuppressants within 2 weeks before the first dose of study therapy;
* (Arm 2 only) Has received a live vaccine within 4 weeks before first dose of study therapy, or potential to receive a live vaccine during the trial treatment;
* Other conditions that might influence the study and analysis of results in the opinion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
ORR by investigator | At baseline, at the time point of every 6 weeks
  ORR is the percentage of evaluable patients with a confirmed investigator-assessed response of CR (complete response) or PR (partial response) per RECIST v1.1 and will be evaluated at baseline, at the time point of every 6 weeks.

SECONDARY OUTCOMES:
DCR by investigator | At baseline, at the time point of every 6 weeks
  DCR is the percentage of evaluable patients with a confirmed investigator-assessed response of CR (complete response), PR (partial response) or SD (stable disease) per RECIST v1.1 and will be evaluated at baseline, at the time point of every 6 weeks.
DoR | up to 2 years
  DoR is the time from the date of first detection of objective response (which is subsequently confirmed) until the date of objective radiographic disease progression.
PFS | up to 2 years
  PFS is the time from the date of first dose until the date of objective radiographic disease progression or death (by any cause in the absence of progression).
OS | up to 2 years
  OS is the time from the date of first dose until the date of death by any cause.
Percentage of participants who experience an adverse event [Safety and Tolerability] | From time of informed consent provided to 3 months after the last dose of study therapy
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. Percentage of participants who experienced an adverse event and discontinued study drug due to an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Hongxia Wang, Chief physician, Principal Investigator — Fudan University; Xichun Hu, Chief physician, Principal Investigator — Fudan University
Locations (1):
- Fudan Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No